CLINICAL TRIAL: NCT06347627
Title: Communicating Human Papillomavirus Vaccine With Japanese Parents and Caregivers With Daughters Aged 12-18: a Mixed-methods Assessment of Acceptance of HPV Vaccine With Experiments on Communication Strategies
Brief Title: Communicating Human Papillomavirus Vaccine With Japanese Parents and Caregivers With Daughters Aged 12-18
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: London School of Hygiene and Tropical Medicine (Other); Nagasaki University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Health Services Research
Other Study IDs: UW23139
Record Dates: First submitted 2024-03-17; First posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-03

CONDITIONS: Healthy
Keywords: HPV Vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (16):
- Group 1 (I x S x S x F) (Experimental): Participants in Group 1 will view a message in an X (former Twitter) format composed of "Individual x Safety x Storytelling x Factual" factors. The message will be available for participants to view while answering five questions that evaluate how it influenced caregivers' trust, confidence, and motivation to vaccinate.
  Interventions: Behavioral: Group 1 (I x S x S x F)
- Group 2 (O x S x S x F) (Experimental): Participants in Group 2 will view a message in an X (former Twitter) format composed of "Organization x Safety x Storytelling x Factual" factors. The message will be available for participants to view while answering five questions that evaluate how it influenced caregivers' trust, confidence, and motivation to vaccinate.
  Interventions: Behavioral: Group 2 (O x S x S x F)
- Group 3 (I x E x S x F) (Experimental): Participants in Group 3 will view a message in an X (former Twitter) format composed of "Individual x Effectiveness x Storytelling x Factual" factors. The message will be available for participants to view while answering five questions that evaluate how it influenced caregivers' trust, confidence, and motivation to vaccinate.
  Interventions: Behavioral: Group 3 (I x E x S x F)
- Group 4 (O x E x S x F) (Experimental): Participants in Group 4 will view a message in an X (former Twitter) format composed of "Organization x Effectiveness x Storytelling x Factual" factors. The message will be available for participants to view while answering five questions that evaluate how it influenced caregivers' trust, confidence, and motivation to vaccinate.
  Interventions: Behavioral: Group 4 (O x E x S x F)
- Group 5 (I x S x S x M) (Experimental): Participants in Group 5 will view a message in an X (former Twitter) format composed of "Individual x Safety x Storytelling x Misinformation" factors. The message will be available for participants to view while answering five questions that evaluate how it influenced caregivers' trust, confidence, and motivation to vaccinate.
  Interventions: Behavioral: Group 5 (I x S x S x M)
- Group 6 (O x S x S x M) (Experimental): Participants in Group 6 will view a message in an X (former Twitter) format composed of "Organization x Safety x Storytelling x Misinformation" factors. The message will be available for participants to view while answering five questions that evaluate how it influenced caregivers' trust, confidence, and motivation to vaccinate.
  Interventions: Behavioral: Group 6 (O x S x S x M)
- Group 7 (I x E x S x M) (Experimental): Participants in Group 7 will view a message in an X (former Twitter) format composed of "Individual x Effectiveness x Storytelling x Misinformation" factors. The message will be available for participants to view while answering five questions that evaluate how it influenced caregivers' trust, confidence, and motivation to vaccinate.
  Interventions: Behavioral: Group 7 (I x E x S x M)
- Group 8 (O x E x S x M) (Experimental): Participants in Group 8 will view a message in an X (former Twitter) format composed of "Organization x Effectiveness x Storytelling x Misinformation" factors. The message will be available for participants to view while answering five questions that evaluate how it influenced caregivers' trust, confidence, and motivation to vaccinate.
  Interventions: Behavioral: Group 8 (O x E x S x M)
- Group 9 (I x S x D x F) (Experimental): Participants in Group 9 will view a message in an X (former Twitter) format composed of "Individual x Safety x Scientific data x Factual" factors. The message will be available for participants to view while answering five questions that evaluate how it influenced caregivers' trust, confidence, and motivation to vaccinate.
  Interventions: Behavioral: Group 9 (I x S x D x F)
- Group 10 (O x S x D x F) (Experimental): Participants in Group 10 will view a message in an X (former Twitter) format composed of "Organization x Safety x Scientific data x Factual" factors. The message will be available for participants to view while answering five questions that evaluate how it influenced caregivers' trust, confidence, and motivation to vaccinate.
  Interventions: Behavioral: Group 10 (O x S x D x F)
- Group 11 (I x E x D x F) (Experimental): Participants in Group 11 will view a message in an X (former Twitter) format composed of "Individual x Effectiveness x Scientific data x Factual" factors. The message will be available for participants to view while answering five questions that evaluate how it influenced caregivers' trust, confidence, and motivation to vaccinate.
  Interventions: Behavioral: Group 11 (I x E x D x F)
- Group 12 (O x E x D x F) (Experimental): Participants in Group 12 will view a message in an X (former Twitter) format composed of "Organization x Effectiveness x Scientific data x Factual" factors. The message will be available for participants to view while answering five questions that evaluate how it influenced caregivers' trust, confidence, and motivation to vaccinate.
  Interventions: Behavioral: Group 12 (O x E x D x F)
- Group 13 (I x S x D x M) (Experimental): Participants in Group 13 will view a message in an X (former Twitter) format composed of "Individual x Safety x Scientific data x Misinformation" factors. The message will be available for participants to view while answering five questions that evaluate how it influenced caregivers' trust, confidence, and motivation to vaccinate.
  Interventions: Behavioral: Group 13 (I x S x D x M)
- Group 14 (O x S x D x M) (Experimental): Participants in Group 14 will view a message in an X (former Twitter) format composed of "Organization x Safety x Scientific data x Misinformation" factors. The message will be available for participants to view while answering five questions that evaluate how it influenced caregivers' trust, confidence, and motivation to vaccinate.
  Interventions: Behavioral: Group 14 (O x S x D x M)
- Group 15 (I x E x D x M) (Experimental): Participants in Group 15 will view a message in an X (former Twitter) format composed of "Individual x Effectiveness x Scientific data x Misinformation" factors. The message will be available for participants to view while answering five questions that evaluate how it influenced caregivers' trust, confidence, and motivation to vaccinate.
  Interventions: Behavioral: Group 15 (I x E x D x M)
- Group 16 (O x E x D x M) (Experimental): Participants in Group 16 will view a message in an X (former Twitter) format composed of "Organization x Effectiveness x Scientific data x Misinformation" factors. The message will be available for participants to view while answering five questions that evaluate how it influenced caregivers' trust, confidence, and motivation to vaccinate.
  Interventions: Behavioral: Group 16 (O x E x D x M)

INTERVENTIONS:
Behavioral: Group 1 (I x S x S x F) — Experimental message: Individual x Safety x Storytelling x Factual
  Arms: Group 1 (I x S x S x F)
Behavioral: Group 2 (O x S x S x F) — Experimental message: Organization x Safety x Storytelling x Factual
  Arms: Group 2 (O x S x S x F)
Behavioral: Group 3 (I x E x S x F) — Experimental message: Individual x Effectiveness x Storytelling x Factual
  Arms: Group 3 (I x E x S x F)
Behavioral: Group 4 (O x E x S x F) — Experimental message: Organization x Effectiveness x Storytelling x Factual
  Arms: Group 4 (O x E x S x F)
Behavioral: Group 5 (I x S x S x M) — Experimental message: Individual x Safety x Storytelling x Misinformation
  Arms: Group 5 (I x S x S x M)
Behavioral: Group 6 (O x S x S x M) — Experimental message: Organization x Safety x Storytelling x Misinformation
  Arms: Group 6 (O x S x S x M)
Behavioral: Group 7 (I x E x S x M) — Experimental message: Individual x Effectiveness x Storytelling x Misinformation
  Arms: Group 7 (I x E x S x M)
Behavioral: Group 8 (O x E x S x M) — Experimental message: Organization x Effectiveness x Storytelling x Misinformation
  Arms: Group 8 (O x E x S x M)
Behavioral: Group 9 (I x S x D x F) — Experimental message: Individual x Safety x Scientific data x Factual
  Arms: Group 9 (I x S x D x F)
Behavioral: Group 10 (O x S x D x F) — Experimental message: Organization x Safety x Scientific data x Factual
  Arms: Group 10 (O x S x D x F)
Behavioral: Group 11 (I x E x D x F) — Experimental message: Individual x Effectiveness x Scientific data x Factual
  Arms: Group 11 (I x E x D x F)
Behavioral: Group 12 (O x E x D x F) — Experimental message: Organization x Effectiveness x Scientific data x Factual
  Arms: Group 12 (O x E x D x F)
Behavioral: Group 13 (I x S x D x M) — Experimental message: Individual x Safety x Scientific data x Misinformation
  Arms: Group 13 (I x S x D x M)
Behavioral: Group 14 (O x S x D x M) — Experimental message: Organization x Safety x Scientific data x Misinformation
  Arms: Group 14 (O x S x D x M)
Behavioral: Group 15 (I x E x D x M) — Experimental message: Individual x Effectiveness x Scientific data x Misinformation
  Arms: Group 15 (I x E x D x M)
Behavioral: Group 16 (O x E x D x M) — Experimental message: Organization x Effectiveness x Scientific data x Misinformation
  Arms: Group 16 (O x E x D x M)

SUMMARY:
This study aims to comprehensively assess confidence in and acceptance of human papillomavirus (HPV) vaccines among Japanese parents and caregivers with daughters aged 12-18 and their decision-making process.

DETAILED DESCRIPTION:
This study will implement an experiment as a sixteen-arm randomized controlled trial in an online survey environment. Before the experiment, participants, who are Japanese caregivers with daughters aged 12-18 who have not received an HPV vaccine, will first answer a pre-experiment survey. The survey will collect information on participants' socio-demographic data and key decision-making factors for HPV vaccine acceptance and confidence. Then, the study will randomly assign the participants to view one digital communication message using a 2 × 2 × 2 × 2 between-person factorial experiment on 'components of message.' The sixteen experimental messages will be developed based on real social media messages posted between November 2021 and April 2022, when the Japanese government prepared to reinstate an active recommendation of HPV vaccines for eligible girls after eight and a half years of suspension.

The sixteen messages will assess four factors: messenger, style, content, and misinformation. Each message will be similar except for one variable in consideration. The messenger component will be whether the message is from an individual or an organization. As individual messengers, the study will set a fictional male or female with common Japanese names who actively communicate about HPV vaccines. As organizational messengers, the study will use the existing accounts of the Ministry of Health, Labour and Welfare or the Japan Cancer Society or a fictional account of an anti-vaccine group. The style component will be whether the message conveys information through storytelling or scientific data. Messages will include personal stories for the storytelling style and statistics for the scientific data style. The content component will be whether the message conveys information about the effectiveness of the HPV vaccine in preventing diseases or the safety of the HPV vaccine. The contents will be built on both factual information and misconceptions about HPV vaccine safety and effectiveness that are often mentioned in the actual social media posts. The misinformation component will be whether the message conveys misinformation or factual information. The study will debrief all respondents exposed to misinformation after the survey.

Lastly, the study will collect data as a post-experiment survey to evaluate how an online message influenced caregivers' trust, confidence, and motivation to vaccinate.

ELIGIBILITY:
Inclusion Criteria:

* Female adult caregivers, older than 20, with daughters aged 12-18 who have received none or only one shot of HPV vaccine.

Exclusion Criteria:

* Caregivers who do not agree to participate in survey, experiment, or both.
* Caregivers with daughters who have already received two or more HPV vaccines.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1600 (Estimated)
Dates: Start 2023-12-22 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Willingness to receive HPV vaccines for daughters | This experiment is expected to take 20-30 minutes to complete. The study will assess the outcome measure immediately after participants are exposed to the experimental messages.
  A degree of a change in willingness to receive HPV vaccines after viewing an experimental message will be scored on a 5-point scale. The options are 1) much less willing to get the HPV vaccine for my daughter, 2) somewhat less, 3) neither more or less, 4) somewhat more, and 5) much more, with higher scores indicating a better outcome.

SECONDARY OUTCOMES:
Confidence in HPV vaccine safety | This experiment is expected to take 20-30 minutes to complete. The study will assess the outcome measure immediately after participants are exposed to the experimental messages.
  A degree of a change in confidence regarding HPV vaccine safety after viewing an experimental message will be scored on a 5-point scale. The options are 1) much less confident that the HPV vaccine is safe, 2) somewhat less, 3) neither more or less, 4) somewhat more, and 5) much more, with higher scores indicating a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Leesa Lin, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- London School of Hygiene and Tropical Medicine, London, United Kingdom

REFERENCES:
- [Derived] Kobayashi K, Masuda K, Wu JT, Lin L. Impact of digital communication message on HPV vaccine decision-making among Japanese mothers: A randomized controlled trial. Vaccine. 2025 Aug 13;61:127327. doi: 10.1016/j.vaccine.2025.127327. Epub 2025 Jun 3. PMID 40466485